CLINICAL TRIAL: NCT02554214
Title: Pilot Clinical Trial on a New Adjustable Glaucoma Drainage Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rheon Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1007
Record Dates: First submitted 2015-09-10; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

ARMS (1):
- Glafkos device (Experimental)
  Interventions: Device: Glafkos drainage device

INTERVENTIONS:
Device: Glafkos drainage device
  Other Names: eyeWatch

SUMMARY:
This will be a prospective, descriptive, mono-center, non-comparative study. A sample of 30 patients who satisfy entry criteria is estimated to be appropriate to provide safety and performance data for this study.

The objectives of the study are to verify the performance and safety of the Glafkos adjustable glaucoma drainage device system. Performance will be measured assessing the possibility to adjust the intra-ocular pressure post-operatively. Safety will be measured by the incidence and severity of adverse events.

The Glafkos device will be implanted in combination with a seton tube. The implant is placed under a scleral flap, in a manner analogous to the ex-Press device (Alcon). The distal end of the draining tube is linked to a seton draining tube, which is linked to a plate placed under the extraocular muscles, creating a filtering space at the orbit (filtering bleb).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or older.
2. Patient shall suffer from primary open angle glaucoma, pseudo-exfoliative glaucoma, or refractory glaucoma after failed previous filtering surgery, in the study eye. Diagnosis is based on glaucomatous optic neuropathy, Shaffer angle greater than 2 as seen on gonioscopy, and visual field defect attributed to glaucoma.
3. Eye to be treated shall be phakic or pseudophakic with no other active ocular disease or disorder except for incipiens cataract. Prior ophthalmic surgery in the study eye shall have been performed more than 3 months before enrollment in this study.
4. Patient condition is indicated for primary and secondary filtration surgery.
5. Presence of ocular hypertension defined as an intraocular corrected pressure (IOP) > 20 mmHg in the study eye, under maximally tolerated medications. The IOP level shall be obtained on 2 consecutive measurements (not taken on the same day) prior to surgery.
6. Distance Snellen best corrected visual acuity (BCVA) better than 0.6 in the fellow eye.
7. For the first three subjects the Snellen BCVA in the study eye should be 0.5 or less. In addition, the visual field defined by the Mean Defect (MD) shall be higher than 10 dB.
8. Optic neuropathy is exclusively attributed to glaucoma.
9. Patient agreed to sign the written inform consent prior to entering into the investigation.
10. Patient is able and willing to complete post-operative follow-up requirements.

Exclusion Criteria:

1. Diagnosis of neovascular glaucoma, congenital glaucoma.
2. History of previous intraocular surgery in the study eye referring to but not limited to extraocular muscles (strabismus), corneal transplant, retinal surgery.
3. Proliferative or severe non-proliferative retinopathy in either eye.
4. Congenital anomaly of the anterior chamber angle in the study eye.
5. Optic neuropathy other than glaucoma in the study eye.
6. Patient with retinal vein occlusion in the study eye.
7. Patient with retinal artery occlusion in the study eye.
8. Patient with corneal opacifications or irregularities that may interfere with the optic nerve evaluation or the IOP measurements in the study eye.
9. Patient with a history of severe eye trauma in the study eye.
10. Patient with ocular malformations such as microphthalmia in the study eye.
11. Patient with concurrent inflammatory/infective eye disorder in the study eye.
12. Patient with any sign of past or present uveitis (anterior/posterior).
13. Patient with severe systemic disease or disabling conditions such as chronic renal failure, post organ transplants.
14. Patient participating in another clinical trial or having participated in another clinical trial less than 3 months prior to entering into the investigation.
15. Patient is pregnant, breast-feeding or unable to make the decision to participate in a clinical investigation (e.g. mentally ill person, mentally handicapped person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number and type of SADE per patient. | 24 months
IOP measurement | 24 months
  IOP reduced by ≥ 20% or IOP < 21 mmHg, and no IOP < 5 mmHg on two consecutive visits after 3 months.

SECONDARY OUTCOMES:
Comprehensive biomicroscopy examination | day 1, day 7, day 14, day 28, month 2, month 3, month 6, month 12, month 18 and month 24
  Anterior and posterior segments examination using a slit-lamp biomicroscope to evaluate the condition of the cornea (epithelium, stroma, endothelium), the anterior chamber, the iris, the lens, the irido-corneal angle (cf. gonioscopy outcome 9), the vitreous body, retinal and optic nerve anatomy (cf funduscopy outcome 7).
Assessment of easiness of surgery by surgeon | day 0
  scale: 0=very easy to 5=very difficult
Assessment of easiness of adjustment | for 24 months
  scale: 0=very easy to 5=very difficult
Subjective refraction | day 7, day 14, day 28, month 2, month 3, month 6, month 12, month 18 and month 24
  Assessment of the subjective refraction based on trial and error asking using trial lenses to achieve the best corrected visual acuity
Funduscopy evaluation | day 7, day 14, day 28, month 2, month 3, month 6, month 12, month 18 and month 24
  indirect funduscopy using a 90D lens to evaluate the optic nerve anatomy (cup to disk ratio measurement) and the retinal structures
Snellen BCVA | day 7, day 14, day 28, month 2, month 3, month 6, month 12, month 18 and month 24
  Distance (6m) decimal visual acuity after best optical correction was provided
gonioscopy assessment | day 7 and day 28
  Irido-corneal angle assessment using the Schaffer grading scale (1-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Montchoisi Clinic, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Roy S, Mermoud A. Efficacy and Safety of an Adjustable Glaucoma Drainage Device (eyeWatch System) for Refractory Glaucoma: A 2-Year Prospective Study. J Glaucoma. 2024 Feb 1;33(2):132-138. doi: 10.1097/IJG.0000000000002334. Epub 2023 Nov 3. PMID 37974333